CLINICAL TRIAL: NCT03021343
Title: Effect of ColchiciNe on the InciDence of Atrial Fibrillation in Open Heart Surgery Patients: END-AF Trial
Brief Title: Effect of Colchicine on the Incidence of Atrial Fibrillation in Open Heart Surgery Patients
Acronym: END-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMC-JCC
Record Dates: First submitted 2015-12-22; First posted 2017-01-13 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Arrhythmia
Keywords: Atrial fibrillation; Colchicine; Cardiac surgery
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Active Comparator): Colchicine 2 mg 12-24 hours prior to surgery and 1 mg 4 hours before or immediately after surgery and then continued at a dose of 0.5 mg twice daily until hospital discharge. Half the dose was given to patients weighing <70 kg or intolerant to the full dose.
  Interventions: Drug: Colchicine
- No colchicine (No Intervention): In this arm no active medication was administered

INTERVENTIONS:
Drug: Colchicine — colchicine given as per trial protocol
  Arms: Colchicine

SUMMARY:
This study evaluates the role of colchicine in the prevention of atrial fibrillation in patients undergoing open heart surgery. Half of participants will receive colchicine and the other half will not

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia in patients undergoing cardiac surgery and is estimated to occur in 26% of all cardiac surgery patients. It can lead to increase morbidity, mainly due to hemodynamic instability and thromboembolic complications, and to increased hospital stay with its associated higher health care cost.

Previous studies have demonstrated that increased inflammation may precede AF and, therefore, interventions that reduce the inflammatory process may help reduce the incidence of AF. Colchicine has potent anti-inflammatory properties and may therefore be capable of reducing the incidence of AF.

This study aims to determine whether the administration of colchicine starting the day before cardiac surgery and continuing until discharge may lead to reduction in post-operative AF.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients undergoing elective cardiac surgery

Exclusion Criteria:

* Documented history of AF or supraventricular arrhythmia or, absence of sinus rhythm on hospital admission
* Known severe liver disease or current transaminases >1.5 times the upper normal limit
* Current serum creatinine >2.5 mg/dl
* Known myopathy or elevated baseline preoperative creatine kinase
* Known blood dyscrasias
* Significant gastrointestinal disease
* Pregnant and lactating women
* Known hypersensitivity to colchicine
* Current treatment with colchicine for any indications
* Emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi A Tabbalat, MD, FACC, Principal Investigator — Khalidi Hospital and Medical Center

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol
Time Frame: 2 years from publication date
Access Criteria: For research purposes after direct contact with principal investigator

REFERENCES:
- [Result] Tabbalat RA, Hamad NM, Alhaddad IA, Hammoudeh A, Akasheh BF, Khader Y. Effect of ColchiciNe on the InciDence of Atrial Fibrillation in Open Heart Surgery Patients: END-AF Trial. Am Heart J. 2016 Aug;178:102-7. doi: 10.1016/j.ahj.2016.05.006. Epub 2016 May 17. PMID 27502857

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colchicine | No Colchicine
Started | 179 | 181
Completed | 174 | 174
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine | No Colchicine | Total
Number analyzed (Participants) | 179 | 181 | 360
Age, Continuous [Mean (Full Range); unit: years] | 60.8 [20 to 82] | 60.5 [23 to 98] | 60.6 [20 to 98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 141 | 143 | 284
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Atrial Fibrillation
Description: The primary efficacy end point was the rate of AF in both arms. AF lasting more than 5 minutes were considered significant
Time Frame: From date of randomization until the date of discharge, assessed up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | No Colchicine
Number analyzed (Participants) | 179 | 181
Participants | 26 | 37

2. Primary Outcome: The Number of Participants With Colchicine Side Effects
Description: The primary safety endpoint was the occurrence of side effects. Side effects monitored were mainly gastrointestinal effects (especially diarrhoea), alopecia, anorexia, hepatotoxicity, myotoxicity, and bone marrow toxicity.
Time Frame: From date of randomization until the date of discharge, assessed up to 2 weeks
Measure: Number; unit: participants
Arm/Group | Colchicine | No Colchicine
Number analyzed (Participants) | 179 | 181
participants | 55 | 14

ADVERSE EVENTS:
Arm/Group | Colchicine | No Colchicine
Serious Adverse Events (participants affected / at risk) | 44/179 | 10/181
Other Adverse Events (participants affected / at risk) | 11/179 | 4/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine (N=179) | No Colchicine (N=181)
Diarrhea (Gastrointestinal disorders) | 44 (44) | 10 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine (N=179) | No Colchicine (N=181)
Anorexia (Gastrointestinal disorders) | 11 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No